CLINICAL TRIAL: NCT01767623
Title: An Open Label, Phase I Study to Evaluate the Impact of Severe Hepatic Impairment on the Pharmacokinetics and Safety of Vemurafenib in BRAF V600 Mutation Positive Cancer Patients
Brief Title: A Study of The Impact of Severe Hepatic Impairment on the Pharmacokinetics and Safety of Vemurafenib in BRAF V600 Mutation-Positive Cancer Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO28053; 2012-003820-18 (EudraCT Number)
Record Dates: First submitted 2013-01-11; First posted 2013-01-14 (Estimated); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — Vemurafenib

ARMS (2):
- Cohort 1: Participants with Normal Liver Function (Active Comparator): Participants with normal liver function (according to National Cancer Institute [NCI] liver dysfunction criteria) will receive vemurafenib 960 mg BID from Day 1 until the morning dose on Day 20 and then from Day 27 onward until disease progression, safety-related treatment termination, withdrawal of consent, death, or a decision by the Sponsor to terminate the study, whichever occurs first.
  Interventions: Drug: Vemurafenib
- Cohort 2: Participants with Severe Liver Dysfunction (Experimental): Participants with severe liver dysfunction (according to NCI liver dysfunction criteria) will receive vemurafenib 720 mg BID from Day 1 until the morning dose on Day 20 and then from Day 27 onward until disease progression, safety-related treatment termination, withdrawal of consent, death, or a decision by the Sponsor to terminate the study, whichever occurs first.
  Interventions: Drug: Vemurafenib

INTERVENTIONS:
Drug: Vemurafenib — Vemurafenib orally BID 960 or 720 mg.
  Other Names: RO5185426; Zelboraf®

SUMMARY:
This open-label, Phase I study will evaluate the impact of severe hepatic impairment on the pharmacokinetics and safety of vemurafenib in participants with BRAF V600 mutation positive cancer. Participants will receive vemurafenib 960 milligrams (mg) (normal hepatic function) or 720 mg (severe hepatic impairment) orally twice daily (BID) on Days 1 to 20 (morning dose) and from Day 27 onward until disease progression or unacceptable toxicity occurs.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed BRAF V600 mutation-positive advanced solid malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective
* Normal or impaired hepatic function (hepatic function will be classified according to the NCI Organ Dysfunction Working Group criteria)
* For participants with hepatic impairment: Stable hepatic function for at least 2 weeks (greater than [>] 14 days) before Day 1
* Eastern Cooperative Oncology Group (ECOG) performance status of less than or equal to (</=) 2
* Participants with a history of recent brain metastases must have completed any radiation therapy at least 4 weeks before Day 1, be without intervening signs of brain lesion progression and not require steroids before starting the protocol (Day 1). Participants with gliomas or known brain metastases who require anticonvulsants must be seizure free for 1 month prior to enrollment
* Life expectancy greater than or eual to (>/=) 8 weeks
* Adequate hematologic and renal function
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of less than (<) 1 percent per year during the treatment period and for at least 6 months after the last dose of study drug

Exclusion Criteria:

* Allergy or hypersensitivity to components of the vemurafenib formulation
* Requirement for immediate or urgent treatment with twice a day vemurafenib and for whom the intermittent schedule of vemurafenib employed during Days 1-26 of this trial is not clinically acceptable
* Chemotherapy, biologic therapy, immunotherapy, or radiotherapy within 4 weeks prior to entering the study, or those who have not recovered from AEs because of agents administered more than 4 weeks earlier
* Gliomas or known brain metastases that require corticosteroids
* History of clinically significant cardiac or pulmonary dysfunction
* Human Immunodeficiency Virus (HIV)-positive participant requiring antiviral treatment including protease inhibitors
* Active infection or chronic infection requiring chronic suppressive antibiotics
* Pregnancy or breastfeeding at Day 1
* History of malabsorption or other clinically significant metabolic dysfunction
* Active autoimmune disease
* Current, recent (within 28 days prior to Day 1), or planned use of any investigational product outside this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-08-20 (Actual); Primary Completion 2017-04-20 (Actual); Study Completion 2017-04-20 (Actual)

PRIMARY OUTCOMES:
Dose-Normalized Area Under the Concentration-Time Curve (AUC) of Vemurafenib During the Dose Interval (12 hours) (AUCtau) on Day 20 | Pre-dose (0 hour); 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, and 168 hours after the morning dose on Day 20
Dose-Normalized Maximum Observed Concentration (Cmax) of Vemurafenib on Day 20 | Pre-dose (0 hour); 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, and 168 hours after the morning dose on Day 20

SECONDARY OUTCOMES:
Percentage of Participants with Adverse Events (AEs) | Baseline up to approximately 3 years
Dose-Normalized AUCtau of of Vemurafenib on Day 1 | Pre-dose (0 hour); 1, 2, 3, 4, 6, 8, and 12 hours after the morning dose on Day 1
Dose-Normalized AUC from Time 0 to Last Measurable Concentration Time Point (AUC0-last) of Vemurafenib on Day 20 | Pre-dose (0 hour); 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, and 168 hours after the morning dose on Day 20
Dose-Normalized AUC from Time 0 to Infinity (AUC0-∞) of Vemurafenib on Day 20 | Pre-dose (0 hour); 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, and 168 hours after the morning dose on Day 20
Dose-Normalized Cmax of Vemurafenib on Day 1 | Pre-dose (0 hour); 1, 2, 3, 4, 6, 8, and 12 hours after the morning dose on Day 1
Time to Maximum Concentration (tmax) of Vemurafenib on Day 1 and Day 20 | Day 1: Pre-dose (0 hour); 1, 2, 3, 4, 6, 8, and 12 hours after the morning dose; Day 20: Pre-dose (0 hour); 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, and 168 hours after the morning dose
Half-life (t1/2) of Vemurafenib in Plasma on Day 20 | Pre-dose (0 hour); 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, and 168 hours after the morning dose on Day 20
Dose Normalized Apparent Clearance (CL/F) of Vemurafenib on Day 20 | Pre-dose (0 hour); 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, and 168 hours after the morning dose on Day 20
Trough Plasma Concentration (Cmin or Ctrough) of Vemurafenib | Pre-dose (0 hour); 1, 2, 3, 4, 6, 8, and 12 hours after the morning dose on Day 1; Pre-dose (0 hour); 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, and 168 hours after the morning dose on Day 20; Before the morning dose on Days 9 and 15

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (8):
- California Cancer Associates for Research & Excellence, Inc., Encinitas, California, United States
- Peninsula and South Eastern Haematology and Oncology Grou, Frankston, Victoria, Australia
- District General Hospital of Athens Laiko; 1st Internal Medicine Clinic, Athens, Greece
- Israel (2):
  - Rambam Health Care Campus, Haifa
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- SBIH " Clinical Oncological Dispensary # 1"; Chemotherapy department #1 and #2, Krasnodar, Russia
- Ege University Medicine Develoment and Pharmacokinetics Research Center; Pulmonary Diseases, Izmir, Turkey (Türkiye)
- Velindre Cancer Centre, Cardiff, United Kingdom